CLINICAL TRIAL: NCT02704975
Title: Effectiveness of Trigger Point Dry Needling and Physical Therapy Versus Physical Therapy Alone Following Shoulder Stabilization Repair: A Randomized Controlled Trial
Brief Title: Effectiveness of Dry Needling and Physical Therapy Versus Physical Therapy Alone Following Shoulder Stabilization Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keller Army Community Hospital (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 16-007
Record Dates: First submitted 2016-03-01; First posted 2016-03-10 (Estimated); Results first posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Shoulder Pain
Keywords: Dry Needling, Shoulder Stabilization
MeSH Terms: conditions — Shoulder Pain | interventions — Rehabilitation; Dry Needling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rehabilitation and Dry Needling (Experimental): Standard Rehabilitation Protocol following shoulder stabilization surgery and Dry Needling to the Shoulder girdle 1 time a week for 4 weeks between weeks 4 and 8 post operatively
  Interventions: Device: Rehabilitation and Dry Needling
- Rehabilitation (Active Comparator): Standard Rehabilitation Protocol following shoulder stabilization surgery alone
  Interventions: Device: Rehabilitation

INTERVENTIONS:
Device: Rehabilitation and Dry Needling — Subjects will receive post-operative rehabilitation that is the standard of care for the surgical procedure they underwent. Rehabilitation will begin within one week after surgery and will continue for the duration of their recovery; two to three treatments a week for approximately 6-9 months. Subjects in this group will also receive dry needling as an adjunct intervention. Dry needling treatment will be performed one time a week for four weeks and will begin four weeks post-operative.
  Arms: Rehabilitation and Dry Needling
Device: Rehabilitation — Subjects will receive post-operative rehabilitation that is the standard of care for the surgical procedure they underwent. Rehabilitation will begin within one week after surgery and will continue for the duration of their recovery; two to three treatments a week for approximately 6-9 months.
  Arms: Rehabilitation

SUMMARY:
The purpose of this single-blinded, randomized clinical trial is to determine the effectiveness of dry needling compared to a standard shoulder rehabilitation program on range of motion, functional movement, and pain in patients who have undergone shoulder stabilization surgery. Measurements of the aforementioned dependent variables will be taken at time intervals of four weeks, eight weeks, 12 weeks, and six months post-operatively. It is hypothesized that the inclusion of dry needling will result in an increase in range of motion, increase in functional movement, and decrease in pain at an accelerated rate when compared to rehabilitation alone.

DETAILED DESCRIPTION:
Methodology /Technical Approach 30-50 subjects at least four weeks after shoulder stabilization surgery will be randomized into two groups (one experimental group and one control group). Subjects in the experimental group will receive Trigger Point Dry Needling (TDN) intervention with standard rehabilitation protocol (Appendix A) while subjects in the control group will receive the same standard rehabilitation protocol without TDN. The experimental group will receive trigger point dry needling one time per week for four to six weeks in addition to the standard rehabilitation protocol. The control group will receive only the standard rehabilitation protocol. Baseline measurements will be taken at approximately four weeks post operatively, and subsequent measurements will be recorded at eight weeks, 12 weeks, and six months.

All patients who have undergone a shoulder stabilization procedure will be invited to participate. Description of the study and informed consent will take place prior to randomization. Concealed randomization will take place 0-7 days post-operatively.

At 4 weeks post-operatively, the following assessment tests will be undertaken: supine shoulder flexion, supine shoulder external rotation, supine shoulder internal rotation, functional movement testing, functional outcome measures, and the numeric pain rating scale. 1,2,3 Those subjects in the 'experimental group' will receive manual palpation of all upper quarter muscles, including the cervical and thoracic spine region, to detect the presence of myofascial trigger points (TPs). Dry needling will be performed to all detected TPs by a provider trained and experienced in TDN.

In addition to the TDN intervention, the experimental group subjects will undergo a rehabilitation program in accordance with a shoulder stabilization repair protocol which is the standard of care for this surgical procedure. Per the shoulder stabilization protocol, subjects will be instructed in a home exercise plan (HEP) that will reinforce the clinical treatment, will be provided with a handout of instructions, and will be required to demonstrate all exercises correctly.

Subjects in the 'control group' will undergo a rehabilitation program as described above for the 'experimental group', except that they will not receive a TDN intervention.

Objectives:

1. To determine if the addition of upper quarter TDN to a rehabilitation protocol is more effective in improving range of motion and functional movement when compared to a rehabilitation protocol alone after shoulder stabilization surgery.
2. To determine if the addition of upper quarter TDN to a rehabilitation protocol is more effective in decreasing pain than a rehabilitation protocol alone after shoulder stabilization surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 yo DOD Beneficiaries
* Status Post Shoulder Stabilization Repair Surgery

Exclusion Criteria:

* Self-Reported Pregnancy
* History of blood borne pathogens/infectious disease/active infection/metal allergy
* Bleeding disorders or currently taking anti-coagulant medications
* Participants who are not fluent in English

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2016-03; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rehabilitation and Dry Needling | Rehabilitation
Started | 19 | 20
Completed | 17 | 19
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rehabilitation and Dry Needling | Rehabilitation | Total
Number analyzed (Participants) | 19 | 20 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] — Age of subjects in years.
  years | 19.9 (1.1) | 21.6 (4.5) | 20.78 (3.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 16 | 17 | 33
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 20 | 39
Numeric Pain Rating Scale (NPRS) [Mean (Standard Deviation); unit: units on a scale] — Numeric Pain Rating Scale. Numerical Scale from 1-10. Subjects are asked self-report pain on a scale from 1 - 10, 1 being the least amount of pain and 10 being the most. The Minimum Important Difference for the NPRS (on a scale from 0-10) range from -1.5 (small change) to -3.0 (medium change) to -3.5 (large change)
  units on a scale | 2.21 (1.8) | 2.55 (1.8) | 2.38 (1.8)
Shoulder Flexion Passive Range of Motion (PROM) [Mean (Standard Deviation); unit: degrees] — Subject is supine with hips and knees flexed for stabilization. Elbow will be extended, forearm relaxed, and wrist in neutral position. Subjects' arm will be raised into forward flexion by the practitioner. The stationary arm of the goniometer will be placed parallel to the spine but at the lateral aspect of the body. The moving arm of the goniometer will be placed along the midline of the humerus.
  degrees | 134.2 (15.1) | 128 (14.5) | 131.1 (14.7)
Shoulder External Rotation (ER) PROM [Mean (Standard Deviation); unit: degrees] — Subject is supine on the plinth with hips and knees flexed for stabilization. Tested arm abducted to 90 degrees. Elbow flexed to 90 degrees. Forearm in the midposition between supination and pronation and perpendicular to the plinth. Subject arm rotated by the practitioner. The stationary arm of the goniometer will be horizontal to the plinth with the pivot of the protractor on the olecranon process. The moving arm of the goniometer is in line with the styloid process of the ulna.
  degrees | 30 (15.9) | 28.67 (21.4) | 29.34 (18.7)
Shoulder Internal Rotation (IR) PROM [Mean (Standard Deviation); unit: degrees] — Subject is supine on the plinth with hips and knees flexed for stabilization. Tested arm abducted to 90 degrees, elbow flexed to 90 degrees, forearm in the midposition between supination and pronation and perpendicular to the plinth,. Subject arm internally rotated by practitioner. Stationary arm of goniometer horizontal to the plinth with the pivot of the protractor on the olecranon process. Moving arm of the goniometer in line with the styloid process of the ulna.
  degrees | 44.5 (12.6) | 36.8 (17.9) | 40.1 (15.6)
Global Rating of Change (GROC) [Mean (Standard Deviation); unit: units on a scale] — Score is rated from -7 (very great deal worse) to +7 (very great deal better) where subjects check an answer that best describes their current perceived status since injury onset to time of follow up. Meaningful patient improvement/deterioration (on a 15 point scale) is considered to be >5 or <-5.
  units on a scale | 4.5 (2) | 4.8 (2) | 4.6 (2)
Shoulder Pain and Disability Index (SPADI) [Mean (Standard Deviation); unit: units on a scale] — The SPADI is a self-report questionnaire assessing pain and disability. The Minimum Important Difference for the SPADI (on a 100- point scale) is 13.2. The total score is reported. Minimum score is 0.
  units on a scale | 42.8 (21.9) | 41.4 (17) | 42 (18.4)
Patient Specific Functional Scale (PSFS) [Mean (Standard Deviation); unit: units on a scale] — The PSFS is a self-report questionnaire assessing pain, instability and activities of daily living (ADLs). The Minimum Important Difference for the PSFS (on a scale from 0-10) range from 1.3 (small change) to 2.3 (medium change) to 2.7 (large change). The total score is reported.
  units on a scale | 2.9 (2.2) | 3.5 (2.1) | 3.2 (2.2)

OUTCOME MEASURES:

1. Primary Outcome: Shoulder Flexion Passive Range of Movement (PROM)
Description: Subject is supine with hips and knees flexed for stabilization. Elbow will be extended, forearm relaxed, and wrist in neutral position. Subjects' arm will be raised into forward flexion by the practitioner. The stationary arm of the goniometer will be placed parallel to the spine but at the lateral aspect of the body. The moving arm of the goniometer will be placed along the midline of the humerus.
Time Frame: at 8 weeks post-op, 12 weeks post-op, 6 months post-op
Population: 3 subjects lost to follow-up between 8 weeks and 6 months. Rows are indicative of multiple timepoints of data collection.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Rehabilitation and Dry Needling | Rehabilitation
Number analyzed (Participants) | 19 | 20
degrees
  8 weeks post-op | 153.9 (12.40) | 153.2 (15.60)
  12 weeks post-op | 164.5 (12.70) | 165.2 (12.30)
  6 months post-op: number analyzed (Participants) | 17 | 19
  6 months post-op | 171.02 (11.49) | 178.7 (4.66)

2. Primary Outcome: Shoulder External Rotation PROM at 8 Weeks
Description: Subject is supine on the plinth with hips and knees flexed for stabilization. Tested arm abducted to 90 degrees. Elbow flexed to 90 degrees. Forearm in the midposition between supination and pronation and perpendicular to the plinth. Subject arm rotated by the practitioner. The stationary arm of the goniometer will be horizontal to the plinth with the pivot of the protractor on the olecranon process. The moving arm of the goniometer is in line with the styloid process of the ulna.
Time Frame: at 8 weeks post-op, 12 weeks post-op, 6 months post-op
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Rehabilitation and Dry Needling | Rehabilitation
Number analyzed (Participants) | 19 | 20
degrees
  8 weeks post-op | 50.05 (17.00) | 51.50 (18.8)
  12 weeks post-op | 64.4 (14.30) | 66.0 (13.8)
  6 months post-op: number analyzed (Participants) | 17 | 19
  6 months post-op | 77.97 (16.32) | 82.13 (12.21)

3. Primary Outcome: Shoulder Internal Rotation (IR) PROM
Description: Subject is supine on the plinth with hips and knees flexed for stabilization. Tested arm abducted to 90 degrees, elbow flexed to 90 degrees, forearm in the midposition between supination and pronation and perpendicular to the plinth,. Subject arm internally rotated by practitioner. Stationary arm of goniometer horizontal to the plinth with the pivot of the protractor on the olecranon process. Moving arm of the goniometer in line with the styloid process of the ulna.
Time Frame: at 8 weeks post-op, 12 weeks post-op, 6 months post-op
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Rehabilitation and Dry Needling | Rehabilitation
Number analyzed (Participants) | 19 | 20
degrees
  8 weeks post-op | 57.3 (11.36) | 55 (15.44)
  12 weeks post-op | 68.9 (10.3) | 63.8 (9.6)
  6 months post-op: number analyzed (Participants) | 17 | 19
  6 months post-op | 71.92 (10.29) | 66.13 (12.64)

4. Secondary Outcome: Global Rating of Change
Description: Score is rated from -7 (very great deal worse) to +7 (very great deal better) where subjects check an answer that best describes their current perceived status since injury onset to time of follow up. Meaningful patient improvement/deterioration (on a 15 point scale) is considered to be >5 or <-5.
Time Frame: at 8 weeks post-op, 12 weeks post-op, 6 months post-op
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rehabilitation and Dry Needling | Rehabilitation
Number analyzed (Participants) | 19 | 20
units on a scale
  8 weeks post-op | 5.32 (1.29) | 5.50 (1.53)
  12 weeks post-op | 5.58 (2.14) | 5.95 (1.09)
  6 months post-op: number analyzed (Participants) | 17 | 19
  6 months post-op | 5.48 (2.72) | 6.6 (0.60)

5. Primary Outcome: Numeric Pain Rating Scale (NPRS)
Description: Numeric Pain Rating Scale. Numerical Scale from 1-10. Subjects are asked self-report pain on a scale from 1 - 10, 1 being the least amount of pain and 10 being the most. The Minimum Important Difference for the NPRS (on a scale from 0-10) range from -1.5 (small change) to -3.0 (medium change) to -3.5 (large change)
Time Frame: at 8 weeks post-op, 12 weeks post-op, 6 months post-op
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rehabilitation and Dry Needling | Rehabilitation
Number analyzed (Participants) | 19 | 20
units on a scale
  8 weeks post-op | 2.2 (1.71) | 1.8 (1.87)
  12 weeks post-op | 1.07 (1.54) | 1.45 (2.04)
  6 months post-op: number analyzed (Participants) | 17 | 19
  6 months post-op | 1.52 (2.17) | 0.90 (1.65)

6. Secondary Outcome: Patient Specific Functional Scale
Description: The PSFS is a self-report questionnaire assessing pain, instability and activities of daily living (ADLs). The Minimum Important Difference for the PSFS (on a scale from 0-10) range from 1.3 (small change) to 2.3 (medium change) to 2.7 (large change). The total score is reported.
Time Frame: at 8 weeks post-op, 12 weeks post-op, 6 months post-op
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rehabilitation and Dry Needling | Rehabilitation
Number analyzed (Participants) | 19 | 20
units on a scale
  8 weeks post-op | 5.78 (2.69) | 6.47 (2.69)
  12 weeks post-op | 6.91 (2.71) | 7.79 (2.42)
  6 months post-op: number analyzed (Participants) | 17 | 19
  6 months post-op | 8.63 (2.09) | 9.21 (1.66)

7. Secondary Outcome: Shoulder Pain and Disability Index Functional Outcome Measure
Description: The SPADI is a self-report questionnaire assessing pain and disability. The Minimum Important Difference for the SPADI (on a 100- point scale) is 13.2. The total score is reported. Minimum score is 0.
Time Frame: at 8 weeks post-op, 12 weeks post-op, 6 months post-op
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rehabilitation and Dry Needling | Rehabilitation
Number analyzed (Participants) | 19 | 20
units on a scale
  8 weeks post-op | 19.3 (16.92) | 18.1 (13.79)
  12 weeks post-op | 10.87 (13.00) | 8.0 (7.01)
  6 months post-op: number analyzed (Participants) | 17 | 19
  6 months post-op | 6.29 (9.83) | 1.96 (1.83)

ADVERSE EVENTS:
Time Frame: 14 months
Description: No serious adverse events were anticipated during this study; there was no all-cause mortality risk in this study. There were no adverse events reported.
Arm/Group | Rehabilitation and Dry Needling | Rehabilitation
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 0/19 | 0/20

LIMITATIONS AND CAVEATS:
There may have been differences in manual therapy received between the two groups. The control group received additional rehab. The follow-up period was also relatively short, at 6 months. The inclusion criteria were also very specific to the subset of the population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-21): https://cdn.clinicaltrials.gov/large-docs/75/NCT02704975/Prot_SAP_000.pdf